CLINICAL TRIAL: NCT00783107
Title: Clinical Investigation of Aerosol Immunotherapy in COPD: A Phase I Placebo-Controlled Dose Escalation/Deescalation Trial of Aerosol Cyclosporine (CyIS) in Patients With Gold Stage III Chronic Obstructive Pulmonary Disease
Brief Title: Aerosol Cyclosporine in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0611109
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Gold Stage III COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine (Experimental)
  Interventions: Drug: Cyclosporine
- Placebo (Placebo Comparator): Subjects will be randomly assigned to Cyclosporine or placebo, in a ratio of 2:1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine — Cyclosporine Inhalation Solution, Once Daily
  Arms: Cyclosporine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, Phase I dose escalation-deescalation protocol (DEP) of cyclosporine inhalation solution in patients with Gold Stage III chronic obstructive pulmonary disease.

The purpose of the study is to evaluate the safety and effectiveness of aerosolized Cyclosporine in treating COPD.

The specific aims of the study are:

1. To identify the short term (28 day) safety profile of CyIS immunotherapy in severe COPD (GOLD III) patients with particular attention to airway reactivity and infection risk.
2. To identify the pharmacokinetic-pharmacodynamic relationship of CyIS using peripheral blood markers of an adaptive immune response as endpoints in subjects with severe COPD (GOLD III) treated short-term.

Subjects between 45 and 70 years of age with a confirmed diagnosis of COPD, Gold Stage III, and meet all the study requirements, will be enrolled in this study. A total of 24 subjects of either sex will be enrolled in this study. A total of 4 subject cohorts (n=6) will participate in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 70 years.
* A confirmed diagnosis of COPD, Gold Stage III, using current accepted diagnostic criteria, including clinical/laboratory findings, pulmonary function tests, and appropriate history to exclude other disorders that could explain their lung disease.
* Subjects agree to maintain a stable medication regimen in the absence of a disease flare
* ECOG performance status of 0, 1, or 2.
* pCO2 < 45 mm Hg, room air oxyhemoglobin saturation > 85%
* A willingness to participate in all portions of the protocol, including serial bronchoscopy, requisite surveillances, and ancillary immunologic studies in follow-up visits at this institution.
* For woman of childbearing age, a negative pregnancy test, and a willingness to use two methods of contraception, or abstinence, and undergo monthly pregnancy testing.
* Elevated T-cell cytokine gene expression, defined as baseline values > the mean of the pilot Gold 0-1 study population for one variable (CD4+IL-2 >23%, CD8+IFN-g >17%, CD8+MHC > 6%, or CD8 TGF-b).
* An ability and willingness to provide written informed consent.

Exclusion Criteria:

* Three, or more exacerbations of lower respiratory disease in the past year requiring systemic corticosteroids, or one exacerbation requiring hospitalization in the past 6 months
* Intubation for COPD, or other cause of respiratory failure in the past year
* Use of immunosuppressive therapy (including oral prednisone), other than aerosolized corticosteroids, anytime within three months prior to participation
* Evidence for an opportunistic infection/colonization of the airways, i.e., non-bacterial
* Use of aerosolized corticosteroids with an inability to maintain inhaled corticosteroid therapy dosing without change during the study interval
* Evidence for systemic illness including hematologic disorders (defined by an absolute neutrophil count (ANC) < 4000 /mL and platelets < 120,000/mL), renal insufficiency (serum creatinine > 2.0 mg/dL), cirrhosis, or hepatic insufficiency (total bilirubin, or alkaline phosphatase > 1.5 x normal, SGOT, or SGPT > 1.2 x normal values), or a coagulopathy (INR > 1.4), seizure disorder.
* Evidence for systemic abnormal renal function manifested by uncontrolled hypertension (systolic blood pressure > 160mmHg or diastolic blood pressure >90mmHg), hyperkalemia (serum creatinine > 5.0 meq/dl, and/or elevated serum creatinine above the normal range for the subject's age.
* Evidence of coronary artery disease by history, e.g., angina or history of myocardial infarction within the past 12 months, unless corrected by CABG within < 5 years, and asymptomatic since
* Pregnant or breast feeding females or women of childbearing potential not practicing birth control during and for 6 months following treatment, or fertile and sexually active males unwilling to use contraceptive techniques during and for 6 months following treatment
* Positive HIV, or hepatitis B or C serology, or another active infection
* Current or past history of cancer excluding basal or squamous cell skin cancer
* Undiagnosed pulmonary nodule requiring diagnostic evaluation
* Weight loss > 10% usual body weight over the past 6 months or a BMI < 18
* Known hypersensitivity or allergy to propylene glycol, CsA, or lidocaine
* Concurrent enrollment or participation within the prior month in other clinical trials
* Greater than 15% or 200 ml reduction in FEV1 post test dose propylene glycol administration
* Known medical or psychological condition (severe personality disorder or mental illness) that would not permit the subject to complete the trial or sign informed consent
* Autoimmune disorders or other disorders with suspected systemic immune involvement
* Active smoking history or urinary cotinine > 2.
* Hypersensitivity to midazolam or narcotics which would not allow bronchoscopy sedation

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and effectiveness of aerosol cyclosporine (CyIS) an immunomodulating therapeutic in treating COPD | Short term (28 day) safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donahoe, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States